CLINICAL TRIAL: NCT00448643
Title: A Phase I Study Using Abdominal Radiotherapy as a Cisplatin Chemosensitizer for Optimally Debulked Stage III/IV Carcinoma of the Endometrium
Brief Title: Whole-Abdominal Radiation Therapy and Cisplatin in Treating Patients With Stage III or Stage IV Endometrial Cancer That Has Been Removed by Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20020138; SCCC-2001064; WIRB-20050721
Record Dates: First submitted 2007-03-15; First posted 2007-03-19 (Estimated); Last update posted 2016-12-15 (Estimated); Status verified 2016-12

CONDITIONS: Endometrial Cancer
Keywords: endometrial adenocarcinoma; endometrial clear cell carcinoma; endometrial papillary carcinoma; stage III endometrial carcinoma; stage IV endometrial carcinoma
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Cisplatin; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Whole-Abdominal Radiation Therapy and Chemotherapy (Experimental)
  Interventions: Radiation: Vaginal Brachytherapy; Drug: Cisplatin; Radiation: Whole Abdominal Radiation [WAR] Therapy

INTERVENTIONS:
Radiation: Vaginal Brachytherapy — High-Dose Rate [HDR] or Low-Dose Rate [LDR], no earlier than during last cycle of Carboplatin/Taxol chemotherapy; or no later than 1 week before cisplation and WAR therapy
Drug: Cisplatin — Weekly at 40 mg/m2 (maximum of 70 mg) for 6 weeks, start no later than 6 weeks from last cycle of standard of care carboplatin and taxol chemotherapy
Radiation: Whole Abdominal Radiation [WAR] Therapy — Whole Abdominal Radiation Therapy, Dose Escalated [2-Levels]; 6 -8 hours after administration of Cisplatin chemotherapy
  Other Names: WAR

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Radiation therapy may also make tumor cells more sensitive to cisplatin. Giving radiation therapy together with cisplatin after surgery may kill any tumor cells that remain after surgery.

PURPOSE: This phase I trial is studying the side effects and best dose of whole-abdominal radiation therapy when given together with cisplatin in treating patients with stage III or stage IV endometrial cancer that has been removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine a recommended phase II dose of adjuvant whole-abdominal radiotherapy when administered with cisplatin in patients with optimally debulked stage III or IV carcinoma of the endometrium.

OUTLINE: This is a dose-escalation study of whole-abdominal radiotherapy (WAR).

Patients receive 3 courses of standard chemotherapy comprising carboplatin IV and paclitaxel IV. Beginning within 6 weeks after completion of standard chemotherapy, patients receive cisplatin IV over 30-60 minutes and undergo a single fraction of WAR on day 1. Treatment with cisplatin and WAR repeats weekly for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Patients may undergo standard vaginal brachytherapy beginning no earlier than the last course of standard chemotherapy or no later than 1 week before the start of cisplatin and WAR.

Cohorts of 3-6 patients receive escalating doses of WAR until the recommended phase II dose (RPTD) is determined. The RPTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. At least 6 patients are treated at the RPTD.

After completion of study treatment, patients are followed periodically.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of endometrial cancer, including any of the following cellular types:

  * Papillary serous carcinoma
  * Clear cell carcinoma
  * Adenocarcinoma
* Stage III or IV disease

  * No evidence of extra-abdominal extension of disease (e.g., groin nodes, lung, or supraclavicular nodes)
* Has undergone total-abdominal hysterectomy, surgical removal of any present fallopian tube and ovary, and resection of any palpable lymph nodes in the pelvis and para-aortic region (or surgical sampling of these nodal regions if no palpable nodes were present) within the past 6 weeks

  * Peritoneal washings must have been collected for cytological evaluation
  * Must have ≤ 1 cm residual disease after surgery

PATIENT CHARACTERISTICS:

* Karnofsky performance status 60-100%
* Life expectancy ≥ 6 months
* WBC ≥ 3,000/mm^3
* Granulocyte count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Creatinine < 2.0 mg/dL
* Bilirubin < 1.5 times upper limit of normal (ULN)
* Lactate dehydrogenase < 3 times ULN
* Gamma glutamyl transferase < 3 times ULN
* SGPT and SGOT < 3 times ULN
* Alkaline phosphatase < 3 times ULN
* No other malignant tumor within the past 5 years

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior radiotherapy to the whole abdomen and/or pelvis/vagina
* No systemic chemotherapy within the past 5 years

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2002-05; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Toxicity as assessed by GOG Common Toxicity Criteria | Study duration
Recommended phase II dose of whole-abdominal radiotherapy | Study duration

CONTACTS AND LOCATIONS:
Overall Officials: Aaron H. Wolfson, MD, Study Chair — University of Miami Sylvester Comprehensive Cancer Center
Locations (1):
- University of Miami Sylvester Comprehensive Cancer Center - Miami, Miami, Florida, United States